CLINICAL TRIAL: NCT04128527
Title: Prospective Non-interventional Evaluation of Insertion and Sealing Performance of AuraOnce Disposable Laryngeal Mask US Version
Brief Title: AuraOnce Performance Observation
Status: Completed | Type: Observational
Sponsor: Ambu A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CIS-016
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Placement of laryngeal mask — All participants are experienced in placement of laryngeal masks and placement will be performed according to standard clinical practice.

SUMMARY:
This study is designed as a single-center, prospective observational, non-controlled, non-interventional study with an investigation period lasting for one day (during one bronchoscopy procedure). The study will take place in Denmark.

The study will include minimum 15 and maximum 20 adult patients planned for a diagnostic flexible bronchoscopy procedure in general anaesthesia using a laryngeal mask. The involved site will include subjects during a one month period, October 2019.

The intention is to perform a quality assessment of the AuraOnce. Subjects will not be asked to participate in this study as it is a quality study where the AuraOnce is used within its intended use and according to normal clinical procedure.

DETAILED DESCRIPTION:
This study is designed as a single-center, prospective observational, non-controlled, non-interventional study with an investigation period lasting for one day (during one bronchoscopy procedure). The study will take place in Denmark.

The study will include minimum 15 and maximum 20 adult patients planned for a diagnostic flexible bronchoscopy procedure in general anaesthesia using a laryngeal mask. The involved site will include subjects during a one month period, October 2019.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years
* Subjects planned for diagnostic flexible bronchoscopy procedure in general anesthesia using a laryngeal mask.

Exclusion Criteria:

- Subjects where use of AuraOnce cannot be clinically justified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for a diagnostic flexible bronchoscopy procedure in general anaesthesia using a laryngeal mask.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults, Laryngeal Mask: Adult patients already scheduled for a diagnostic flexible bronchoscopy procedure in general anesthesia using a laryngeal mask.
Period: Overall Study
Arm/Group | Adults, Laryngeal Mask
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No baseline data was collected on participants
Groups:
- Adults, Laryngeal Mask: Adult patients (> 18 years) already scheduled for a diagnostic flexible bronchoscopy procedure in general anesthesia using a laryngeal mask.
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 0
Age, Continuous [unit: years] — Population: Continuous Age Data were not collected
Sex: Female, Male — Sex/gender data were not collected Population: Sex/Gender data were not collected
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Leakage Observed During Procedure
Description: Is leakage observed (yes/no) if yes, insert signs of leakage
Time Frame: During procedure, less than 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 16
Participants | 0

2. Secondary Outcome: Investigator Evaluation of Ease of Insertion on a 5-point Scale (Very Difficult (=1) to Very Easy (=5))
Description: Investigator evaluation of ease of insertion on a 5-point scale (very difficult (=1) to very easy (=5))
Time Frame: During procedure, less than 1 hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 16
score on a scale | 4.6 (0.7)

3. Secondary Outcome: Investigator Evaluation of Ease of Obtaining Seal on a 5-point Scale (Very Difficult (=1) to Very Easy (=5))
Description: Investigator evaluation of ease of obtaining seal on a 5-point scale (very difficult (=1) to very easy (=5))
Time Frame: During procedure, less than 1 hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 16
score on a scale | 4.7 (0.6)

4. Secondary Outcome: Investigator Evaluation of Overall Performance on a 5-point Scale (Very Bad (=1) to Excellent (=5))
Description: Investigator evaluation of overall performance on a 5-point scale (very bad (=1) to excellent (=5))
Time Frame: During procedure, less than 1 hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 16
score on a scale | 4.6 (0.5)

5. Secondary Outcome: Number of Participants With Correct Placement of Mask
Description: It is checked if the mask is placed above the vocal cords (yes/no)
Time Frame: During procedure, less than 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 16
Participants | 16

6. Secondary Outcome: Number of Participants Where Tip of the Mask is Folded
Description: After insertion of the mask, it is assessed by bronchoscopy whether the tip of the mask is folded. Folded tip= Yes, Not folded= No
Time Frame: During procedure, less than one hour
Measure: Count of Participants; unit: Participants
Arm/Group | Adults, Laryngeal Mask
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Time Frame: Data collected over the course of one month, Adverse Events assessed during each procedure (less than 1 hour)
Arm/Group | Adults, Laryngeal Mask
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT04128527/Prot_SAP_000.pdf